CLINICAL TRIAL: NCT04400149
Title: The Effect of Maternal Serum and Amniotic Fluid Progesterone Levels on Pregnancy Results
Brief Title: Progesterone Levels and Pregnancy Results
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Tufan Arslanca, M.D., Ufuk University
Other Study IDs: amniotic fluid progesteron
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy Complications; Pregnancy Preterm; Pregnancy Loss
MeSH Terms: conditions — Pregnancy Complications | interventions — Amniocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: amniotic fluid progesterone (this group will be evaluated by the amniotic fluid which was received via amniocentesis). This group consisted of pregnant women who had high risk in the antenal test and give consent to perform amniocentesis. Notwithstanding, amniocentesis detects chromosome abnormalities, neural tube defects, and genetic disorders for the fetuses. İn a routine amniocentesis, 1-2 ml amniotic fluid which was taken in the first place was discarded in order to prevent maternal contamination. Then 15-20 ml amniotic fluid was taken from all of the patients to diagnose genetic disorders of the fetuses. İn this study we evaluate the amniotic fluid progesterone in this 1-2 ml amniotic fluid which was discarded and throw away. Therefore, we are not performing an extra invasive procedure for pregnant women
  Interventions: Diagnostic Test: amniocentesis
- 2: serum progesterone (this group consisted of the pregnant women who have amniocentesis procedure and blood samples were taken in the same procedure )
  Interventions: Diagnostic Test: amniocentesis

INTERVENTIONS:
Diagnostic Test: amniocentesis — amniocentesis will be performed to the pregnant women at 16-20 weeks who had a high-risk antenatal test. Furthermore, these women also give a blood sample (at 16-20 weeks) to compare the amniotic fluid and serum progesterone levels in association with pregnancy outcomes. We perform amniocentesis to evaluate genetic disorders in pregnant women who had his risk in the antenal test.

SUMMARY:
The aim of this study is to evaluate the amniotic fluid and serum progesterone level and pregnancy outcome

DETAILED DESCRIPTION:
Studies have investigated the relationship between maternal serum progesterone level and low birth weight baby birth, hypertensive disorders of pregnancy, and early pregnancy bleeding. In some cases, patients are supported by oral or vaginal progesterone treatments during pregnancy. We also measure the relationship between maternal serum progesterone by measuring the level of amnion progesterone; We aimed to analyze the effects on pregnancy outcomes by observing preterm birth, premature rupture of membranes, low birth weight, baby gender, maternal problems that may occur during pregnancy, fetal problems.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Women who did not receive progesterone treatment during pregnancy

Exclusion Criteria:

* Women who receive progesterone treatment during pregnancy
* multiple pregnancies
* Diagnosed hypertension, diabetes mellitus, kidney disease, heart disease, liver disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study population consists of 18-45 years old pregnant women who had a high risk in the antenatal screening test and give consent to perform amniocentesis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
pregnancy outcome | starting from 16 weeks, ending at the delivery of the baby
  premature membran rupture Web sonuçları
  Premature Rupture of Membranes
pregnancy outcome | starting from 16 weeks, ending at the delivery of the baby
  pregnancy loss
pregnancy outcome | starting from 16 weeks, ending at the delivery of the baby
  preeclampsia
pregnancy outcome | starting from 16 weeks, ending at the delivery of the baby
  gestational diabetes

SECONDARY OUTCOMES:
fetal outcomes | starting from 16 weeks, ending at the delivery of the baby
  low birth weight
fetal outcomes | starting from 16 weeks, ending at the delivery of the baby
  preterm labor
fetal outcomes | starting from 16 weeks, ending at the delivery of the baby
  fetal gender

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johansson ED, Jonasson LE. Progesterone levels in amniotic fluid and plasma from women. I. Levels during normal pregnancy. Acta Obstet Gynecol Scand. 1971;50(4):339-43. doi: 10.3109/00016347109157335. No abstract available. PMID 5157500
- [Result] Lau IF, Saksena SK, Salmonsen R. The concentration of progesterone, 20 alpha-dihydroprogesterone, testosterone, oestrone and oestradiol-17 beta in serum, amniotic fluid and placental tissue of pregnant rabbits. Acta Endocrinol (Copenh). 1982 Apr;99(4):605-11. doi: 10.1530/acta.0.0990605. PMID 7072456
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Progesterone+levels+in+amniotic+fluid+and+plasma+from+women.+I.+Levels+during+normal+pregnancy
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=The+concentration+of+progesterone%2C+20%5Cg%3Da%5C-dihydroprogesterone%2C+testosterone%2C+oestrone+and+oestradiol-17%5Cg%3Db%5Cin+serum%2C+amniotic+fluid+and+placental+tissue+of+pregnant+rabbits